CLINICAL TRIAL: NCT02259517
Title: Imaging Stimulant vs. Non-Stimulant Treatment of Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: An fMRI Study of Stimulant vs. Non-Stimulant Treatment of ADHD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment/enrollment ended early due to the COVID-19 pandemic
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); American Academy of Child Adolescent Psychiatry. (Other); Shire (Industry)
Responsible Party: Principal Investigator, Jonathan Posner, Associate Professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6961
Record Dates: First submitted 2014-09-30; First posted 2014-10-08 (Estimated); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Intuniv; Non-stimulant; Guanfacine extended-release; Vyvanse; Stimulant; Lisdexamfetamine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guanfacine (Experimental): Participants will be administered extended-release guanfacine, which is in tablet form, and will be instructed to take the medication once daily for 6 weeks. The daily dose will range between 1 and 4 mg.
  Interventions: Drug: Guanfacine
- Lisdexamfetamine (Experimental): Participants will be administered lisdexamfetamine, which is in tablet form, and will be instructed to take the medication daily for 6 weeks. The daily dose will range between 30 and 70mg.
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Guanfacine — Participants will meet with the study doctor on a weekly basis during the treatment phase of the study. In the first few weeks, the daily dose of the medication will be individually adjusted by the study doctor according to participants' clinical response to and tolerability of the medication. The optimal dose will then be maintained for the remainder of the treatment period.
  Other Names: Intuniv; GXR
  Arms: Guanfacine
Drug: Lisdexamfetamine — Participants will meet with the study doctor on a weekly basis during the treatment phase of the study. In the first few weeks, the daily dose of the medication will be individually adjusted by the study doctor according to participants' clinical response to and tolerability of the medication. The optimal dose will then be maintained for the remainder of the treatment period.
  Other Names: Vyvanse; LDX
  Arms: Lisdexamfetamine

SUMMARY:
Children with Attention-Deficit/Hyperactivity Disorder (ADHD) are typically treated with two types of medications with differing mechanisms of action: stimulants and non-stimulants. The stimulant Vyvanse (lisdexamfetamine, LDX), and the non-stimulant Intuniv (extended-release guanfacine, GXR), are both FDA approved treatment for ADHD. Clinical trials have shown that both medications are effective in reducing ADHD symptoms, although the neurobiological mechanisms by which Vyvanse and Intuniv produce these effects remain unknown. The aim of this study is to examine the mechanisms by which LDX and GXR reduce symptoms in patients with ADHD. MRI scanning will be used to identify treatment-related changes in brain structure and function.

DETAILED DESCRIPTION:
Children with ADHD and age and sex-matched healthy controls will be scanned at the beginning of the study. In this first part of the study, MRI findings will be compared between the two groups to see whether brain functioning of children with ADHD differs from that of healthy children. In the second part of the study, the children with ADHD will meet weekly with the study doctor and be administered either extended-release guanfacine (Intuniv) or lisdexamfetamine (Vyvanse) for 6 weeks. Selection into either treatment group will be randomly determined. At the end of the study, the children with ADHD treated with either medication will have a second MRI scan. The findings of that second MRI scan will be compared to the first MRI scan in order to examine brain changes due to the medication. These second MRI scans will also be compared to the scans of the healthy controls.

ELIGIBILITY:
Inclusion Criteria:

ADHD Participants:

* The participant satisfies Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a primary diagnosis of ADHD, any subtype.

Healthy Control Participants:

* The participant must have no current DSM Axis I psychiatric disorder.

All Participants:

* Participants must provide assent and a legal guardian must provide consent.
* The participant is male or female and between 6 - 17 years of age and in good physical health.
* Girls of childbearing potential must have a negative urine pregnancy test and, if sexually active, must be using adequate contraception.
* The participant is English speaking.

Exclusion Criteria:

ADHD Participants:

* The participant has a current comorbid DSM Axis I psychiatric diagnosis or other symptomatic manifestations that, in the opinion of the study doctor, will contraindicate lisdexamfetamine or guanfacine treatment or confound safety assessments.
* The participant meets DSM-5 criteria for current substance abuse and/or dependence.
* The participant is currently taking or has taken within the past 4 months, a psychotropic medication.
* The participant has a documented allergy or intolerance to lisdexamfetamine or guanfacine products.
* The participant has a diagnosis or a history of cardiovascular disease or any other serious medical illness.
* The participant is pregnant or lactating.
* The participant is actively suicidal.
* MRI contraindications (e.g., irremovable metal on the body, pacemaker, braces)
* The participant has a full-scale intelligence quotient (IQ) less than 70.
* The participant has a history of seizure (except febrile seizure).

Healthy Controls:

* The participant meets DSM criteria for current substance abuse and/or dependence.
* The participant is currently taking a psychotropic medication.
* The participant has a history of a serious medical illness.
* The participant is pregnant or lactating.
* MRI contraindications (e.g., irremovable metal on the body, pacemaker, braces)
* The participant has a full-scale intelligence quotient (IQ) less than 70.
* The participant has a history of seizure (except febrile seizure).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Posner, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in 2014 and ended in 2020. Participants were primarily recruited from the community through advertisements in local newspapers and flyers posted in local establishments. Participants were also recruited from other research studies and doctor's offices.
Pre-assignment Details: 5 ADHD participants withdrew or were excluded from the study prior to randomization and thus are not included. Participants who withdrew were no longer interested in treatment or were lost to follow-up. Participants were excluded due to subthreshold ADHD symptoms, comorbid psychiatric conditions, & MRI contraindications.
Groups:
- ADHD - Guanfacine: ADHD participants who were randomized to receive guanfacine for 6 weeks of treatment
- ADHD - Lisdexamfetamine: ADHD participants who were randomized to receive lisdexamfetamine for 6 weeks of treatment
- Healthy Controls: Age- and sex- matched healthy control participants; baseline procedures only
Period: Overall Study
Arm/Group | ADHD - Guanfacine | ADHD - Lisdexamfetamine | Healthy Controls
Started | 5 | 4 | 24
Completed | 5 | 4 | 15
Not Completed | 0 | 0 | 9
Not completed — Psychiatric diagnosis (e.g., ADHD, MDD) | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | ADHD - Guanfacine | ADHD - Lisdexamfetamine | Healthy Controls | Total
Number analyzed (Participants) | 5 | 4 | 15 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (2.35) | 8.75 (0.96) | 9.6 (2.47) | 9.54 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 8 | 10
  Male | 4 | 3 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 5 | 7
  Not Hispanic or Latino | 2 | 1 | 1 | 4
  Unknown or Not Reported | 2 | 2 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 8 | 10
  White | 2 | 2 | 3 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 4 | 6
Behavior Rating Inventory of Executive Function, 2nd Edition - Global Executive Composite [Mean (Standard Deviation); unit: T-score] — The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) assesses executive function in children and adolescents ages 5-18 years old. The Global Executive Composite (GEC) is an overall summary score and reflects all the clinical scales of the BRIEF-2. Higher scores indicate lower levels of executive functioning. Parent-report T-scores on the GEC are reported below (population mean = 50, population standard deviation = 10). Population: One Healthy Control participant was missing the parent-report BRIEF-2.
  T-score
    number analyzed (Participants) | 5 | 4 | 14 | 23
    (all) | 65.33 (7.77) | 62.5 (9.33) | 44.57 (12.38) | 52.22 (14.47)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Segmentation Volume Produced by Stimulant or Non-stimulant Medications in Patients With ADHD
Description: Brain segmentation volume measured in mm^3. We are reporting the mean difference in brain segmentation volume from baseline (pre-test) to 6 weeks (post-test).
  No statistical analysis information is being submitted for the affected outcome measure. No statistical analyses have been performed or would be considered scientifically appropriate because actual enrollment fell well below target enrollment. Enrollment terminated early as a result of the COVID-19 pandemic.
Time Frame: Baseline and 6 weeks
Population: 4 subjects from the ADHD-Guanfacine group and 3 subjects from the ADHD-Lisdexamfetamine group had usable anatomical MRI data at baseline and follow-up. HCs did not complete follow-up.
  No statistical analysis information is being submitted for the affected outcome measure. No statistical analyses have been performed or would be considered scientifically appropriate because actual enrollment fell well below target enrollment. Enrollment terminated early as a result of the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | ADHD - Guanfacine | ADHD - Lisdexamfetamine
Number analyzed (Participants) | 4 | 3
mm^3 | -6137 (14393) | 11833 (39942)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, an average of 6 weeks.
Description: Adverse events were routinely collected from ADHD participants receiving treatment using the Pittsburgh Side Effects Rating Scale. A physician met with participants in person approximately once per week during treatment. The physician was also available by phone between visits.
  HC participants completed a baseline assessment and did not receive any intervention; therefore, there was no monitoring for adverse events.
Arm/Group | Guanfacine | Lisdexamfetamine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
No statistical analysis information is being submitted for the affected outcome measure. No statistical analyses have been performed or would be considered scientifically appropriate because actual enrollment fell well below target enrollment. Enrollment terminated early as a result of the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT02259517/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT02259517/SAP_001.pdf